CLINICAL TRIAL: NCT03894891
Title: Sequential Therapy With Induction TPN Followed by Nivolumab With Radiation in Locoregionally Advanced Laryngeal and Hypopharyngeal Cancer
Brief Title: Induction TPN Followed by Nivolumab With Radiation in Locoregionally Advanced Laryngeal and Hypopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert Haddad, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-652
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; Cisplatin; Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) then Radioimmunotherapy (IMRT+N) then adjuvant N (Experimental): Participants received 3 cycles of induction with docetaxel, cisplatin and nivolumab (TPN) every 3 weeks (or 21 days): docetaxel 75 mg/m2 IV day 1, cisplatin 100 mg/m2 IV day 1, and nivolumab 240 mg IV flat dose day 1.
  Induction was followed by clinical and radiologic assessment of response. Participants without partial response or better based on RECIST 1.1 were offered salvage laryngectomy and/or pharyngectomy. Participants with partial or complete response per RECIST 1.1 proceeded with immunoradiotherapy concurrently with nivolumab. Intensity-modulated radiotherapy (IMRT) was preferred and proton beam radiotherapy not permitted. Nivolumab 240 mg IV flat dose day 1 was repeated every 2 weeks concurrently with IMRT (for a total of 3-4 doses).
  Participants then received adjuvant nivolumab (480 mg IV flat dose day 1) every 4 weeks within 3-8 weeks from the last day of IMRT for up to 6 cycles or until disease progression or recurrence.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a type of immunotherapy.
  Other Names: OPDIVO®
Drug: Cisplatin — Cisplatin is a chemotherapy drug.
  Other Names: Platinol
Drug: Docetaxel — Docetaxel is a chemotherapy drug.
  Other Names: Taxotere
Radiation: Intensity-modulated radiotherapy — IMRT is definitive treatment for head and neck cancer.
  Other Names: IMRT

SUMMARY:
This research is being performed to treat patient for head and neck cancer patients who have not received prior chemotherapy.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug or combination of interventions is being studied.

Nivolumab is approved by the U.S. Food and Drug Administration (FDA) for the treatment of recurrent or advanced head and neck cancer (head and neck cancer that has come back or is incurable) but is considered investigational for head and neck cancer patients who have not received prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically or cytologically confirmed, resectable or unresectable, Stage III or Stage IV locoregionally advanced squamous cell carcinoma of the larynx or hypopharynx, as defined by 2017 American Joint Committee on Cancer (AJCC), 8th edition
* Willing to provide tissue from diagnostic biopsy and blood samples before, during, and after treatment
* Any smoking history is permitted
* Patients must have HPV negative disease. Those patients with a supraglottic primary are required to undergo HPV testing with p16 immunohistochemistry and/or confirmatory HPV PCR or ISH testing to rule out oropharyngeal origin with laryngeal extension
* Age 18 years or older
* ECOG performance status ≤ 1 (Karnofsky ≥ 80%, see Appendix A)
* Participant must have normal organ and marrow function as defined below within 21 days prior to study registration:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤2.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception. WOCBP should plan to use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 iu/l or equivalent units of hcg) within 24 hours prior to the start of nivolumab
* Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

Exclusion Criteria:

* Existing severe autoimmune conditions (at the discretion of the treating physician). Patients with a history of Hashimoto thyroiditis who are stable on replacement hormone therapy are not excluded. Short-term corticosteroid dosing is permitted (i.e. dexamethasone for chemotherapy-induced nausea prevention during induction chemotherapy) as long as steroids are discontinued within 1 week (7 days) of receiving the first dose of nivolumab during the induction phase of treatment.
* Subject who has had prior chemotherapy for head and neck cancer and/or radiotherapy to the head and neck.
* Subject who has been treated with immunotherapy. This includes prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known human immunodeficiency virus carrier or a diagnosis of immunodeficiency. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
* Known non-infectious pneumonitis or any history of interstitial lung disease.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low-risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease in the last 5 years is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Tisch Cancer Institute, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: December 19, 2019 to November 3, 2020
Period: Overall Study
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Started | 6
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Completed protocol treatment per protocol | 5

BASELINE CHARACTERISTICS:
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Laryngectomy-free Survival (LFS)
Description: LFS defined as time from study registration to earlier of surgical removal of larynx and/or hypopharynx, or death due to any cause. Participants alive with intact larynx and hypopharynx are censored at date of last disease evaluation. Given limited sample size and zero events, the Kaplan-Meier method was not used for estimate of LFS.
Time Frame: Disease was assessed following the completion of 2-3 cycles of induction TPN, 10-12 weeks after the completion of immunoradiotherapy or surgery and every 3 months until disease progression (PD). Participants were followed up to 18.9 months.
Measure: Median (Full Range); unit: months
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
months | 11.1 [1.8 to 18.9]

2. Secondary Outcome: Best Radiologic Response
Description: Best radiologic response on treatment was evaluated per RECIST 1.1 criteria. For target lesions: complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Non-CR/Non-PD defined as persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Disease evaluation following the completion of the induction phase of treatment on cycle 3 day 43-63.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
Participants
  Complete Response | 3
  Partial Response | 2
  Non-CR/Non-PD | 1

3. Secondary Outcome: Median Censoring Time for Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from study entry to death or censored at date last known alive. Given limited sample size and zero events, the Kaplan-Meier method was not used for the estimate of OS. The empirical median is provided which represents median time to date last known alive (all 6 participants were censored).
Time Frame: Participants were observed for OS up to 23.2 months.
Measure: Median (Full Range); unit: months
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
months | 12.9 [2.8 to 23.2]

4. Secondary Outcome: Median Laryngo-esophageal Dysfunction-free Survival (LEDFS)
Description: LEDFS is defined as time from study registration to earlier of surgical removal of larynx and/or hypopharynx, non-functioning larynx and/or hypopharynx (inability to swallow, speak, and/or breath on own), or death from any cause. Participants alive with intact and functioning larynx and hypopharynx and esophagus are censored at date of last disease evaluation. Given limited sample size and zero events, the Kaplan-Meier method was not used for estimate of LEDFS.
Time Frame: Disease was assessed following the completion of 2-3 cycles of induction TPN, 10-12 weeks after the completion of immunoradiotherapy or surgery and every 3 months until disease progression (PD). Participants were observed for LEDFS up to 18.9 months.
Measure: Median (Full Range); unit: months
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
months | 11.1 [1.8 to 18.9]

5. Secondary Outcome: EORTC QLQ-C30 Change in Emotional Functional Score From Baseline to Post IMRT+Nivolumab
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. The emotional functional (EF) scale has 3 items (v3 items 21-24). Scores are standardized to range from 0-100. Higher scores indicate better emotional health.
Time Frame: At baseline and post IMRT+Nivolumab approximately 22 weeks from start of induction treatment.
Population: The evaluable population represents participants with the QLQ-C30 completed at both assessment times.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 5
units on a scale | 8.3 [-16.7 to 25.0]

6. Secondary Outcome: Number of Participants With Grade 3-5 Treatment-related Adverse Events
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 The number of treated participants experiencing at least one of these adverse events as defined during the time of observation was counted.
Time Frame: AEs were evaluated up to 9.6 months, representing maximum treatment duration for this study cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 6
Participants | 3

7. Secondary Outcome: EORTC QLQ-C30 Change in Fatigue Score From Baseline to Post IMRT+Nivolumab
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. The fatigue scale has 3 items (v3 items 10,12,18). Scores are standardized to range from 0-100. Higher scores indicate more symptomatology.
Time Frame: At baseline and post IMRT+Nivolumab approximately 22 weeks from start of induction treatment.
Population: The evaluable population represents participants with the QLQ-C30 completed at both assessment times.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Induction Docetaxel (T)+Cisplatin (P)+Nivolumab (N) Then Radioimmunotherapy (IMRT+N) Then Adjuvant N
Number analyzed (Participants) | 5
units on a scale | 33.3 [-33.3 to 66.7]

ADVERSE EVENTS:
Time Frame: AEs were evaluated up to 9.6 months, representing maximum treatment duration for this study cohort. All-cause mortality was evaluated up to 23.2 months, representing maximum survival for this study cohort.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining AEs regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated in these two subsets of data. No further data is available to specify classification of other beyond the general term.
Groups:
- Docetaxel+Cisplatin+Nivolumab+Radioimmunotherapy: Docetaxel will be administered per standard institutional every 3 weeks Nivolumab will be administered intravenously every 3 weeks Cisplatin will be administered intravenously every 3 weeks Radioimmunotherapy will be conducted 3 weeks after the last cycle of TPN (docetaxel, cisplatin and nivolumab)
  Nivolumab: Nivolumab is a type of immunotherapy that tries to enhance participants own immune system to fight cancer
  Cisplatin: Cisplatin is a chemotherapy medication used to treat a number of cancers
  Docetaxel: Docetaxel (Taxotere®) is a chemotherapy drug. It is used to treat many types of cancer including head and neck
  Radioimmunotherapy: Radiation Therapy to shrink or kill tumors.
Arm/Group | Docetaxel+Cisplatin+Nivolumab+Radioimmunotherapy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel+Cisplatin+Nivolumab+Radioimmunotherapy (N=6)
Anemia (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel+Cisplatin+Nivolumab+Radioimmunotherapy (N=6)
Anemia (Blood and lymphatic system disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Infections and infestations - Other (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Investigations - Other (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Serum amylase increased (Investigations) | 2
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study terminated early due to weak accrual and therefore no inference is possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03894891/Prot_SAP_000.pdf